CLINICAL TRIAL: NCT00427128
Title: Prozac Treatment of Major Depression: Discontinuation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4099R; RO1 MH56058
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Major Depression
Keywords: Major Depression; "true drug" response; "placebo response" pattern; continuation treatment outcomes
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: fluoxetine — 10mg/day increased over 12 weeks to 20-80 mg/day; 20-80 mg/day maintained from week 13-36.
  Other Names: Prozac
Drug: placebo — Week 13-36.

SUMMARY:
This study randomized two stratifications of acute phase MDD SSRI responders, categorized as having either "true drug" response or "placebo response" pattern, to continuation with SSRI vs placebo in a double-blind trial to determine if stratification category predicted continuation outcome.

DETAILED DESCRIPTION:
This study enrolled 627 subjects with Major Depressive illness at New York State Psychiatric Institute and Massachusetts General Hospital. Subjects were treated with fluoxetine 10-60mg over a 12 week period. The "responder" group was defined by those no longer meeting criteria for Major Depression at week 12, along with CGI ratings of "much improved" or "very much improved" as determined by an independent evaluator. At week 12 "non-responders" were withdrawn from the study and received open label treatment; responders were randomized in double-blind fashion to either fluoxetine continuation (20-80mg daily) at response dose or placebo switch for up to 24 weeks. The responder group was stratified by "specific or true" drug response (late onset and persistent once attained) and "nonspecific or placebo" response (early onset or nonpersistent) patterns. Subjects were evaluated at one week and two week intervals at different phases of continuation treatment, and depression relapse was determined by agreement between study psychiatrist and independent evaluator CGI and Ham-D ratings, as well as administration of the MDD section of the Mood Disorders Module of the Structured Clinical Interview for DSM-IV Disorders at those visits. A subset of study participants also provided DNA samples to determine whether there are any DNA markers of response type. Data were analyzed to test the following hypotheses: that during continuation fluoxetine treatment improved patients with a "true drug" acute response pattern randomized to placebo had a poorer outcome than those maintained on active drug; that during continuation fluoxetine treatment improved patients with a "placebo" acute response pattern randomized to placebo had no worse an outcome than those maintained on drug; that during continuation fluoxetine treatment patients with a "true drug" acute response pattern randomized to continue on fluoxetine were more likely to maintain their benefit than those with a "placebo" pattern.

ELIGIBILITY:
Inclusion Criteria:

1. men and women ages 18-65
2. meets criteria for DSM IV Major Depression
3. signs informed consent and able to comply with study

Exclusion Criteria:

1. pregnant women and women of child-bearing potential who are not using a medically accepted means of contraception.
2. women taking oral contraceptives, the initiation of which was temporally associated with the onset of depression; women who are breast-feeding.
3. Patients with serious suicidal risk, including any patient who became suicidal with previous discontinuation of an antidepressant.
4. Patients with a history of seizure disorder.
5. Patients with unstable physical disorders (cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic) or any physical disorder judged to significantly affect CNS function.
6. Patients meeting criteria for the following DSM-IV diagnoses: organic mental disorders; substance use disorders, including alcohol, active within the last 6 months; schizophrenia; delusional disorder; psychotic disorders; bipolar disorder; antisocial personality disorder; or presence of psychotic features
7. Patients with a history of non-response to an adequate trial of a selective serotonin reuptake inhibitor in a past or current depressive episode, defined as a four-week trial of a minimum of 40mg/day of fluoxetine or paroxetine, or 100mg/day of sertraline.
8. Concurrent use of exclusionary drugs
9. Clinical or laboratory evidence of hypothyroidism without adequate stable replacement (eg, low total T4 or elevated TSH by a high sensitivity method).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 1995-11; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
MDD section of Mood Disorders Module of Structured Clinical Interview for DSM-IV (SCID) | up to 9 mos.
Ham-D | up to 9 mos.
CGI | up to 9 mos.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McGrath, MD, Principal Investigator — New York State Psychiatric Institute; Maurizio Fava, MD, Principal Investigator — Massachussets General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York State Psychiatric Institute, New York, New York

REFERENCES:
- [Result] McGrath PJ, Stewart JW, Quitkin FM, Chen Y, Alpert JE, Nierenberg AA, Fava M, Cheng J, Petkova E. Predictors of relapse in a prospective study of fluoxetine treatment of major depression. Am J Psychiatry. 2006 Sep;163(9):1542-8. doi: 10.1176/ajp.2006.163.9.1542. PMID 16946178
- [Derived] Posternak MA, Baer L, Nierenberg AA, Fava M. Response rates to fluoxetine in subjects who initially show no improvement. J Clin Psychiatry. 2011 Jul;72(7):949-54. doi: 10.4088/JCP.10m06098. Epub 2011 May 31. PMID 21672502
- [Derived] Yang H, Sinicropi-Yao L, Chuzi S, Youn SJ, Clain A, Baer L, Chen Y, McGrath PJ, Fava M, Papakostas GI. Residual sleep disturbance and risk of relapse during the continuation/maintenance phase treatment of major depressive disorder with the selective serotonin reuptake inhibitor fluoxetine. Ann Gen Psychiatry. 2010 Feb 26;9:10. doi: 10.1186/1744-859X-9-10. PMID 20187924
- See also: official site of Depression Evaluation Service — http://www.depression-nyc.org